CLINICAL TRIAL: NCT00819494
Title: Role of Skin Tests for the Diagnosis of Immediate Hypersensitivity Reactions Due to Iodinated Contrast Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Jettanong Klaewsongkram, MD, Chulalongkorn University
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Chula-ARC 003/08
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Hypersensitivity
Keywords: Contrast media skin test; Skin test; hypersensitivity; contrast media
MeSH Terms: conditions — Hypersensitivity | interventions — Skin Tests; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy controls (Sham Comparator)
  Interventions: Procedure: Skin tests with radiocontrast media
- Patients with immediate reactions (Active Comparator)
  Interventions: Procedure: Skin tests with radiocontrast media

INTERVENTIONS:
Procedure: Skin tests with radiocontrast media — Skin prick tests and intradermal test will be performed in patients with a history of immediate reactions to iodinated radiocontrast media

SUMMARY:
The purpose of this trial is to study the diagnostic role of skin test in immediate reactions to iodinated radiocontrast media.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of immediate hypersensitivity reactions to iodinated contrast media
2. 15-70 years of age

Exclusion Criteria:

1. On antihistamine/ cannot discontinue antihistamine before the test
2. Having asthma exacerbation
3. Being pregnant
4. Suffering from severe systemic disease/ in bad health

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Percentages of positive wheal and flare responses from skin test in patients with a history of immediate reactions to radiocontrast media | 5 months

SECONDARY OUTCOMES:
Blood in vitro test from patients with a history of immediate reactions to radiocontrast media | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand